CLINICAL TRIAL: NCT03427294
Title: Delphi Study on Rehabilitation Following Lumbar Arthrodesis in UZ Leuven (Belgium)
Brief Title: Delphi Study on Rehabilitation Following Lumbar Arthrodesis
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: UHasselt (Unknown); KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: KU/UZ Leuven S60109 - 2
Record Dates: First submitted 2018-01-26; First posted 2018-02-09 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-02

CONDITIONS: Lumbar Spine Degeneration; Physical Disability; Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Care providers involved in lumbar arthrodesis: surgeons, physiotherapists, behavioral therapists, researchers, occupational therapists
  Interventions: Other: Delphi study

INTERVENTIONS:
Other: Delphi study — Delphi study on the optimal rehabilitation pathway following lumbar arthrodesis

SUMMARY:
Delphi study on perioperative rehabilitation after single and double level lumbar arthrodesis.

DETAILED DESCRIPTION:
The investigators aim to engage all care providers in Belgium and the Netherlands who are at some point involved in the rehabilitation path related to single and double level lumbar arthrodesis.

ELIGIBILITY:
Inclusion Criteria:

* The investigators aim to engage all care providers (Belgium, the Netherlands) who are involved in the care of patients following lumbar arthrodesis.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators aim to engage all care providers (Belgium, the Netherlands) who are involved in the care of patients following lumbar arthrodesis.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Duration of perioperative rehabilitation following lumbar arthrodesis | January - December 2018
  duration defined in amount of weeks
Physiotherapeutic content following lumbar arthrodesis | January - December 2018
  describing the physiotherapeutic modalities defined as manual therapy, exercise therapy, or cognitive behavioural therapy
Frequency of physiotherapeutic intervention following lumbar arthrodesis | January - December 2018
  frequency defined as amount of physiotherapeutic visits per week
Multidisciplinary character of perioperative rehabilitation following lumbar arthrodesis | January - December 2018
  amount and type of involved health care providers, as well as the interaction between

CONTACTS AND LOCATIONS:
Overall Officials: Bart Depreitere, PhD, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Thijs Swinnen, MSc, PT, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Tinne Thys, MSc, PT, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Wim Dankaerts, PhD, PT, Principal Investigator — KU Leuven; Simon Brumagne, PhD, PT, Principal Investigator — KU Leuven; Peter Van Wambeke, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Lieven Moke, PhD, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Sebastiaan Schelfaut, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Ann Spriet, MSc, PT, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Lotte Janssens, PhD, PT, Principal Investigator — Hasselt University
Locations (1):
- UZ/KU Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thys T, Bogaert L, Dankaerts W, Depreitere B, Van Wambeke P, Brumangne S, Bultheel M, Vanden Abeele V, Moke L, Spriet A, Schelfaut S, Janssens L, Swinnen TW. Qualitative study exploring the views of patients and healthcare providers on current rehabilitation practices after lumbar fusion surgery. BMJ Open. 2024 May 30;14(5):e077786. doi: 10.1136/bmjopen-2023-077786. PMID 38816040